CLINICAL TRIAL: NCT01576081
Title: The Effects of a 56day Unilateral Muscular Unloading Intervention With a Novel Device That Allows Normal Ambulation While Reducing Muscle Activation Drastically, on Muscles, Bones and Vessels.
Brief Title: The Novel Unloading Device "HEPHAISTOS" and Its Effects Upon Bone, Muscle and Vasculature
Acronym: HEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DLR German Aerospace Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DLR
Record Dates: First submitted 2012-04-03; First posted 2012-04-12 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-08

CONDITIONS: Bone Resorption
Keywords: bone density; weight bearing; muscle atrophy; vascular degeneration; gravitational loading; muscular unloading
MeSH Terms: conditions — Bone Resorption; Muscular Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Unilateral orthotic intervention (Experimental): The HEPHAISTOS orthotic was worn unilaterally for 56days by 11 healthy male subjects.
  Interventions: Device: HEPHAISTOS

INTERVENTIONS:
Device: HEPHAISTOS — HEPHAISTOS unloading orthotic

SUMMARY:
The present study aimed to investigate the importance of gravitational induced forces that appear during normal ambulation for the health of muscles, bones and blood vessels. The main hypothesis of the present study is that gravitational loading alone, without muscle contractions, is insufficient to maintain bone strength.

DETAILED DESCRIPTION:
The 56day unloading intervention with HEPHAISTOS had the following key objectives:

1. Primary objective: Assessment and evaluation of bone adaptation.
2. Secondary objective: Assessment and evaluation of functional and structural muscular adaptations.
3. Third objective: Assessment and evaluation of functional and structural vascular adaptations.
4. Fourth objective: Assessment and evaluation if the present findings deviate from findings observed in established unloading models.

ELIGIBILITY:
Inclusion Criteria:

* male
* age: 20-40 years
* BMI: 20-30
* passing the psychological and medical check up.
* signed consent to participate in the study
* faultless certificate of good conduct

Exclusion Criteria:

* smoking
* professional athletes
* diabetes
* muscle or joint disease
* trabecular bone density in the distal tibia epiphysis < 160mg/cm3
* increase risk of thrombosis
* bone fractures 12 months prior to the study
* metal implants, any material of osteosynthesis
* participation in another clinical intervention study 2 months prior to the study
* bleeding disorder
* anesthetic intolerance
* vascular disease
* epilepsy
* claustrophobia
* herniated disk
* pacemaker
* alcohol or drug abuse
* anti-inflammatory drug intake during the study
* hyperlipidemia
* kidney disease
* hyperhomocysteinaemia
* vitamin d deficit
* chronical back pain
* detained

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2011-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Bone density as measured with pQCT | 1 year
  subjects will be followed for one year, starting from the onset of the study

CONTACTS AND LOCATIONS:
Overall Officials: Joern Rittweger, Prof. Dr., Study Director — DLR German Aerospace Center; Tobias Weber, Principal Investigator — DLR German Aerospace Center; Michel Ducos, Principal Investigator — DLR German Aerospace Center
Locations (1):
- German Aerospace Center, Cologne, Germany

REFERENCES:
- [Derived] Weber T, Ducos M, Mulder E, Beijer A, Herrera F, Zange J, Degens H, Bloch W, Rittweger J. The relationship between exercise-induced muscle fatigue, arterial blood flow and muscle perfusion after 56 days local muscle unloading. Clin Physiol Funct Imaging. 2014 May;34(3):218-29. doi: 10.1111/cpf.12087. Epub 2013 Oct 7. PMID 24119174
- [Derived] Weber T, Ducos M, Mulder E, Herrera F, Bruggemann GP, Bloch W, Rittweger J. The specific role of gravitational accelerations for arterial adaptations. J Appl Physiol (1985). 2013 Feb;114(3):387-93. doi: 10.1152/japplphysiol.01117.2012. Epub 2012 Dec 6. PMID 23221961
- See also: Webpage German Aerospace Center (DLR), Division Space Physiology — http://www.dlr.de/me/desktopdefault.aspx/tabid-1935/